CLINICAL TRIAL: NCT05144386
Title: A Phase 1/2a, Sequential Cohort, Single Ascending Dose Study of the Safety, Tolerability, Biodistribution, and Pharmacodynamics of EBT 101 in Aviremic HIV-1 Infected Adults on Stable Antiretroviral Therapy
Brief Title: Study of EBT-101 in Aviremic HIV-1 Infected Adults on Stable ART
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Excision BioTherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EBT-101-001
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-07

CONDITIONS: HIV-1-infection
Keywords: CRISPR; Gene Therapy; AAV9; HIV; SaCas9

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EBT-101 Dose-Level 1 (Experimental): Cohort A: Participants will be administered dose-level 1 of EBT-101
  Interventions: Biological: EBT-101
- EBT-101 Dose-Level 2 (Experimental): Cohort B: Participants will be administered dose-level 2 of EBT-101
  Interventions: Biological: EBT-101

INTERVENTIONS:
Biological: EBT-101 — EBT-101 is a HIV-1-specific clustered regularly interspaced short palindromic repeats (CRISPR)/Cas9 gene editing system delivered by adenovirus-associated virus vector serotype 9 (AAV9) for intravenous (IV) administration

SUMMARY:
This is a First in Human (FIH) study of EBT-101 administered IV to aviremic HIV-1 infected adults on stable antiretroviral therapy (ART).

DETAILED DESCRIPTION:
This is a FIH, open-label, sequential cohort, single ascending dose (SAD) study of EBT-101 administered IV to aviremic HIV-1 infected adults on stable ART.

Participants will be asked to attend several visits for screening to determine eligibility. On Day 1, eligible participants will receive a single IV dose of EBT-101. All participants will be assessed for eligibility for an analytical treatment interruption (ATI) of their background ART at Week 12. All participants will be followed through Week 48 (end of study). Participants are required to attend multiple study visits at the clinical site including daily visits for the first 14 days, followed by weekly visits after Week 12 for ATI participants. Non-ATI participants are followed monthly after Week 12.

Eligible participants who are enrolled in the FIH study (EBT-101-001) will also be enrolled in a separate Long Term Follow Up (LTFU) study (EBT-101-002) for safety monitoring. The duration of the LTFU study is 15 years.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

* Willing to enroll and sign the written informed consent for EBT-101-001 (current study) and EBT-101-002, the LTFU study.
* Age between 18 and 70 years (both inclusive).
* Weight: Cohort A ≥55 and ≤110 kg, Cohort B ≥55 and ≤90 kg.
* Cohorts A and B will only enroll male subjects (sex at birth).
* Chronic HIV-1 with known subtype B infection
* On stable regimen defined as continuous ART suppressive treatment with HIV RNA level below the level of quantitation for >1 years prior to screening
* Plasma HIV-1 RNA levels below the limit of quantitation during screening.
* Peripheral blood CD4 T cell count ≥500 cells/mm3 for at least 2 years prior to screening
* Willing and able to comply, as assessed by the Investigator, with all study-related procedures.
* Have previously been vaccinated for N. meningitidis with documented history and/or received a N. meningitidis vaccination prior to dosing.
* Willing to stop ART if eligible for analytical treatment interruption.
* Willing to comply with the measures to prevent HIV transmission and reinfection required by the protocol.
* Must have received a COVID-19 vaccination series and boosters as specified by current federal (CDC) recommendations, with the last dose ≥30 days prior to dosing.

Exclusion Criteria (abbreviated):

* Documented prior HIV-1 drug resistance to ≥2 or more classes of ART defined as single key mutations or an accumulation of minor mutations that result in resistance to entire respective drug classes within the past 5 years.
* History of >1 change in ART due to virologic failure during preceding 2 years prior to screening.
* Received in the preceding 12 months or HCP plans to prescribe long-acting injectable ART.
* History of HIV dementia.
* History of progressive multifocal leukoencephalopathy.
* History of significant cardiac disease in last 2 years.
* History of HIV-related kidney disease with abnormal renal function.
* Known history and/or documented: pre-HIV treatment nadir CD4+ T cell count <200 cells/mm3 or post-suppressive HIV treatment confirmed CD4+ T cell <200 cells/mm3 prior to screening
* History of AIDS-defining opportunistic infection prior to screening.
* Evidence of acute or chronic hepatitis B and/or hepatitis C.
* Known history or diagnosis of liver cirrhosis.
* Diagnosis of nonalcoholic fatty liver or advanced nonalcoholic steatohepatitis.
* Predefined abnormal laboratory values within 42 days of dosing per protocol
* Known history of positive tuberculin skin test.
* Receipt of any investigational HIV vaccine (prophylactic and/or therapeutic) within the year prior to screening.
* Receipt of any gene therapy product approved or experimental, at any time.
* Anti-AAV9 serum neutralizing antibodies (Nabs) >1:20 titer.
* Known positive SARS-CoV-2 test within 48 hours prior to planned dosing date.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cohorts A and B will enroll male adults (sex at birth)
Enrollment: 6 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of EBT-101 | 48 weeks
  Safety and tolerability of EBT-101 will be assessed based on the incidence and severity of adverse events (AEs) according to Division of AIDS (DAIDS) 2017 over 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Kennedy, MD, Study Director — Excision BioTherapeutics
Locations (3):
- United States (3):
  - Quest Clinical Research, San Francisco, California
  - Washington University, St Louis, Missouri
  - Cooper Health, Camden, New Jersey

IPD SHARING:
Plan to Share IPD: No